CLINICAL TRIAL: NCT01566929
Title: Weight Management Interventions for Obese Women and the Live Birth Outcome of in Vitro Fertilization (IVF): a Randomized Controlled Trial
Brief Title: Weight Management Intervention for Obese Women and the Live Birth Outcome of in Vitro Fertilization (IVF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Skane University Hospital (Other); Region Örebro County (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other); Herlev Hospital (Other); Holbaek Sygehus (Other); ART Medica clinic, Iceland (Unknown)
Responsible Party: Principal Investigator, Ann Thurin Kjellberg, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Obesity/IVF
Record Dates: First submitted 2012-03-23; First posted 2012-03-30 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Infertility; Obesity
Keywords: Obesity; In vitro fertilization; Low calorie diet (LCD); Obstetric outcome; Weight reduction
MeSH Terms: conditions — Infertility; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVF only (No Intervention): IVFtreatment
- Weight reduction treatment and IVF (Active Comparator): Dietary Supplement: Low calorie diet treatment and then IVFtreatment
  Interventions: Dietary Supplement: Low calorie diet treatment

INTERVENTIONS:
Dietary Supplement: Low calorie diet treatment — Reduction of calorie intake to only 800 kcal/day by using LCD during 12 weeks
  Arms: Weight reduction treatment and IVF

SUMMARY:
The primary aim of the study is to evaluate if weight management intervention for obese women (BMI≥30<35 kg/m2) prior to IVF improves the outcome assessed as live birth per participating woman, as compared to women where no intervention was made.

DETAILED DESCRIPTION:
1. There will be two groups of patients.

   1. The first group (n=167) will receive weight management intervention during up to four months prior to IVF treatment.The group randomized to intervention will start an intensive weight reduction plan. The aim of the weight reduction is to reach as close to normal BMI (<25.0 kg/m2) as possible during a time of approximately 4 months. The purpose of the dietary intervention is to create a negative energy balance to induce weight loss. The intervention starts with 12 weeks of a low calorie liquid formula diet (LCD) and thereafter, diet re-introduction and weight control stabilization until IVF treatment begins. Should the patient for some reason be unable to fulfil the LCD-treatment, she will anyhow have an individualized dietary counselling to help her loose weight until the time for her IVF-treatment.
   2. The second group (n=167) will start their IVF-treatment directly without other intervention than written advice about the benefits of weight reduction and exercise. The group randomized directly to IVF-treatment will start the treatment as soon as possible after randomization, preferably within that menstrual cycle.
2. Tertiary aim is a follow-up 2 years after randomization to the study with questionnaires to the couple in both the intervention and the control groups. A special questionnaire will cover the weights of the couple and if the woman has had any pregnancies or live births after concluding the study. For the women having achieved a live birth in the index-cycle of IVF the number of children and also follow-up of the children will be performed by assessing medical records from pediatric clinic (if applicable) and child health care centres covering birth data, general health and weight of the children at birth and at the assessment date. Eating -habits and -patterns and quality of life parameters will be assessed with the same three questionnaires that were filled in after randomization.

ELIGIBILITY:
Inclusion criteria

* Indication for IVF/ICSI for the couple
* Woman's age >18< 38 years at randomization
* First, second or third IVF/ICSI treatment
* BMI > or = 30.0 <35.0 kg/m2
* Willing to participate and to sign informed consent

Exclusion Criteria:

* Diabetes mellitus treated with insulin
* Oocyte or sperm donation planned
* Preimplantation genetic diagnosis (PGD) treatment planned
* Azoospermia known at randomization
* Patient not having adequate knowledge of Swedish (to understand patient information and questionnaires)
* QEWP-R questionnaire indicating binge eating disorder for the woman
* Previous participation in the study

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 317 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Live birth | Approximately 10-16 months after randomization, depending on study group.
  Live birth per participating woman

SECONDARY OUTCOMES:
embryology | After theIVF-treatment, approximately 1-6 months after randomization
  number of good quality embryos
obstetric outcomes | Approximately 10-16 months after randomization, after delivery
  obstetric and neonatal data
compliance to intervention | Assessed in the intervention group 12-16 weeks after randomization, prior to IVF-treatment
  Compliance to intervention assessed as weight loss during intervention, dietary intake and quality of life
Husband data | before IVF-treatment
  Measurement of the husband for height, weight and dietary intake and eating patterns correlated to sperm count, sperm motility and sperm chromatin fragmentation

CONTACTS AND LOCATIONS:
Overall Officials: Ann Thurin Kjellberg, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (9):
- Denmark (4):
  - Herlev hospital, Copenhagen
  - Hvidovre hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Holbaek hospital, Holbæk
- ART Medica, Reykjavik, Iceland
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes Universitetssjukhus, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska Universitetssjukhuset, Stockholm

REFERENCES:
- [Derived] Svensson H, Einarsson S, Olausson D, Kluge L, Bergh C, Eden S, Lonn M, Thurin-Kjellberg A. Inflammatory and metabolic markers in relation to outcome of in vitro fertilization in a cohort of predominantly overweight and obese women. Sci Rep. 2022 Aug 3;12(1):13331. doi: 10.1038/s41598-022-17612-2. PMID 35922472
- [Derived] Kluge L, Bergh C, Einarsson S, Pinborg A, Mikkelsen Englund AL, Thurin-Kjellberg A. Cumulative live birth rates after weight reduction in obese women scheduled for IVF: follow-up of a randomized controlled trial. Hum Reprod Open. 2019 Dec 10;2019(4):hoz030. doi: 10.1093/hropen/hoz030. eCollection 2019. PMID 31844684
- [Derived] Einarsson S, Bergh C, Friberg B, Pinborg A, Klajnbard A, Karlstrom PO, Kluge L, Larsson I, Loft A, Mikkelsen-Englund AL, Stenlof K, Wistrand A, Thurin-Kjellberg A. Weight reduction intervention for obese infertile women prior to IVF: a randomized controlled trial. Hum Reprod. 2017 Aug 1;32(8):1621-1630. doi: 10.1093/humrep/dex235. PMID 28854592